CLINICAL TRIAL: NCT05598229
Title: To Observe a Multicenter, Randomized, Controlled Clinical Study on the Effect of Tiktok on Perioperative Emotions of Patients Undergoing Bone Prosthesis Replacement
Brief Title: Application of Douyin in Perioperative Period of Malignant Tumor Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZZUSC-14
Record Dates: First submitted 2022-10-23; First posted 2022-10-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-10

CONDITIONS: Malignant Tumor of Bone; Perioperative Period
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watch the Tik Tok (Experimental): Encouraged to watch the Tik Tok.
  Interventions: Other: Tik Tok
- Tik Tok is not allowed (No Intervention): Tik Tok is not allowed.

INTERVENTIONS:
Other: Tik Tok — Encourage and do not restrict watching Tik Tok
  Arms: Watch the Tik Tok

SUMMARY:
Fitting into the group of 90 cases of this study was to henan tumor hospital bone prosthesis replacement of surgical treatment of bone malignant tumors patients, evaluate watch trill to be bone prosthesis replacement surgery treatment of malignant bone tumor patients perioperative anxiety, depression, pain, explore watch trill to bone prosthesis replacement surgery treatment of malignant bone tumor patients of postoperative complications.

DETAILED DESCRIPTION:
Fitting into the group of 90 cases of this study was to henan tumor hospital bone prosthesis replacement of surgical treatment of bone malignant tumors patients, evaluate watch trill to be bone prosthesis replacement surgery treatment of malignant bone tumor patients perioperative anxiety, depression, pain, explore watch trill to bone prosthesis replacement surgery treatment of malignant bone tumor patients of postoperative complications. Eligible subjects were screened and treated with the following treatment regimen: Experimental group: Enrolled patients were encouraged to watch Douyin without limit from 24 hours before surgery to 30 minutes before surgery. He was encouraged to watch Douyin without limit until the seventh day after surgery. Control group: Viewing Douyin was forbidden from 24 hours before enrollment to the seventh day after operation. The Hospital Anxiety and Depression Self-rating Scale (HADS) and Visual analogue Scale (VAS) were used to detect the anxiety and depression of the subjects. 2. Anxiety and depression values 30 minutes before surgery; 3. Anxiety value, depression value and pain value 24 hours after operation. 4. Anxiety value, depression value and pain value at 48 hours after operation. Incidences of surgery-related complications were observed at 1 month after operation.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 10-70. The Eastern Collaborative Oncology Group (ECOG) physical status score was 0-1. Subjects with amputation can be relaxed up to 2 points.

Pathological diagnosis of malignant tumor. Patients undergoing bone prosthesis replacement for bone tumors. All acute toxicities due to previous antitumor therapy or surgery resolved to grade 0-1 (according to NCI-CTCAE version 5.0) or to enrollment/exclusion criteria by day 1 of the first cycle (C1D1), except for toxicities such as hair loss that the investigator considered to pose no safety risk to the subject).

Adequate organ and bone marrow function, as defined below:

Blood routine (no blood transfusion, no G-CSF, no medication correction within 7 days before screening) :

Neutrophil count (ANC)≥1,500/mm3(1.5×109/L); Platelet count (PLT)≥100,000/mm3(100×109/L); Hemoglobin (Hb)≥9g/dL(90g/L);

Blood biochemical:

Serum creatinine (Cr)≤1.5× upper limit of normal (ULN) or creatinine clearance (Cockroft-Gault formula)≥60ml/min; Total bilirubin (TBIL)≤1.5×ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤2.5×ULN, and subjects with liver metastases should ≤5×ULN;

Blood coagulation function:

International normalized ratio (INR)≤1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT)≤1.5×ULN; With my consent and signed informed consent, I am willing and able to comply with the planned visit, study treatment, laboratory tests and other test procedures.

Exclusion Criteria:

Received the following treatment within 14 days before C1D1:

Radiotherapy, chemotherapy, immune or molecularly targeted therapy for tumors. Some other investigational drugs. Surgery for other sites and/or radiotherapy were planned during the study period (24 hours before surgery to 7 days after surgery).

Imaging diagnosis showed the presence of central nervous system tumor lesions. The presence of active heart disease in the 6 months before C1D1, including myocardial infarction, severe/unstable angina pectoris, etc. Poorly controlled arrhythmias with left ventricular ejection fraction <50% on echocardiography (including QTcF interval >450ms in men and >470ms in women).

In the judgment of the investigator, there are concomitant diseases (such as severe diabetes, neurological or psychiatric diseases) or any other conditions that seriously endanger the safety of the subjects, may confuse the results of the study, or affect the completion of the study.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 48 hours before surgery
  A moving scale measuring about 10cm in length was used, with 10 scales on one side and "0" and "10" ends, respectively, with 0 indicating no pain and 10 indicating the most severe pain that could not be endured. In clinical evaluation, "0-2" was classified as "excellent", "3-5" was classified as "good", "6-8" was classified as "fair", and > 8 was classified as "poor".
Hospital Anxiety Depression Scale | 24 hours before surgery
  Two subscales, anxiety and depression, were included. 0-7 were asymptomatic, 8-10 were suspicious, and 11-21 were definitely present.
Hospital Anxiety Depression Scale | 30 minutes before surgery
  Two subscales, anxiety and depression, were included. 0-7 were asymptomatic, 8-10 were suspicious, and 11-21 were definitely present.
Hospital Anxiety Depression Scale | 24 hours after surgery
  Two subscales, anxiety and depression, were included. 0-7 were asymptomatic, 8-10 were suspicious, and 11-21 were definitely present.
Visual Analogue Scale | 24 hours after surgery
  A moving scale measuring about 10cm in length was used, with 10 scales on one side and "0" and "10" ends, respectively, with 0 indicating no pain and 10 indicating the most severe pain that could not be endured. In clinical evaluation, "0-2" was classified as "excellent", "3-5" was classified as "good", "6-8" was classified as "fair", and > 8 was classified as "poor".
Hospital Anxiety Depression Scale | 48 hours after surgery
  Two subscales, anxiety and depression, were included. 0-7 were asymptomatic, 8-10 were suspicious, and 11-21 were definitely present.
Visual Analogue Scale | 48 hours after surgery
  A moving scale measuring about 10cm in length was used, with 10 scales on one side and "0" and "10" ends, respectively, with 0 indicating no pain and 10 indicating the most severe pain that could not be endured. In clinical evaluation, "0-2" was classified as "excellent", "3-5" was classified as "good", "6-8" was classified as "fair", and > 8 was classified as "poor".

IPD SHARING:
Plan to Share IPD: No